CLINICAL TRIAL: NCT00222053
Title: IFM 99-02 Thalidomide in Myeloma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: LLAU ME, University Hospital Toulouse
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PHRC 98-45-N
Record Dates: First submitted 2005-09-15; First posted 2005-09-22 (Estimated); Last update posted 2010-04-02 (Estimated); Status verified 2010-04

CONDITIONS: Multiple Myeloma
Keywords: Myeloma; Autologous transplantation; Maintenance therapy; Thalidomide
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell | interventions — Thalidomide; Diphosphonates

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (No Intervention): No specific intervention
- 2 (Active Comparator): Biphosphonates
  Interventions: Drug: Biphosphonates
- 3 (Experimental): Thalidomide
  Interventions: Drug: Thalidomide

INTERVENTIONS:
Drug: Thalidomide — Per os thalidomide
  Arms: 3
Drug: Biphosphonates — Biphosphonates
  Arms: 2

SUMMARY:
Principal objective is to evaluate the impact of Thalidomide to prolong the duration of response after autologous transplantation for myeloma

ELIGIBILITY:
Inclusion Criteria:

* de novo myeloma
* according to Durie and Salmon classification stage II, III and stage I with a lytic bone lesion
* patients from 18 to 65 years old
* beta2microglobulin < 3 mg/l or del13 absent
* signed informed consent
* eligible for transplantation

Exclusion Criteria:

* peripheral neurological toxicities
* uncontrolled or severe cardiovascular disease
* other malignancy except basocellular carcinoma or FIGO stage I carcinoma of the cervix
* patient who received biphosphonate during the last 60 days
* renal failure definited as creatinine > 150 µmol/l
* patient with obvious vascular cerebral medical history
* liver dysfunction definited as bilirubin > 35 µmol/l or ASAT, ALAT, PAL > 4N
* respiratory dysfunction
* HIV +
* Patient who refused to use an acceptable barrier method for contraception

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Actual)
Dates: Start 2000-04; Primary Completion 2009-09 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Duration of response | 3 years

SECONDARY OUTCOMES:
Survival | 3 years
Toxicity | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: ATTAL Michel, MD, Principal Investigator — University Hospital, Toulouse
Locations (5):
- France (5):
  - Médecine Interne, CHU Purpan, Toulouse
  - Médecine Interne, Hôpital Rangueil, Toulouse
  - Rhumatologie, CHU Purpan, Toulouse
  - Rhumatologie, CHU Rangueil, Toulouse
  - Service d'hématologie, CHU Purpan, Toulouse

REFERENCES:
- [Background] Combination chemotherapy versus melphalan plus prednisone as treatment for multiple myeloma: an overview of 6,633 patients from 27 randomized trials. Myeloma Trialists' Collaborative Group. J Clin Oncol. 1998 Dec;16(12):3832-42. doi: 10.1200/JCO.1998.16.12.3832. PMID 9850028
- [Background] Attal M, Harousseau JL, Stoppa AM, Sotto JJ, Fuzibet JG, Rossi JF, Casassus P, Maisonneuve H, Facon T, Ifrah N, Payen C, Bataille R. A prospective, randomized trial of autologous bone marrow transplantation and chemotherapy in multiple myeloma. Intergroupe Francais du Myelome. N Engl J Med. 1996 Jul 11;335(2):91-7. doi: 10.1056/NEJM199607113350204. PMID 8649495